CLINICAL TRIAL: NCT01214460
Title: Impact of Medical Emergency Team and EMS on ICU Readmissions and Sudden Cardiac Arrests in Tampere University Hospital
Brief Title: Impact of Medical Emergency Team and EMS in Tampere University Hospital
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R10111
Record Dates: First submitted 2010-07-05; First posted 2010-10-05 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Death, Sudden,Cardiac
Keywords: MET
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- All MET calls: We make an Utstein type analyze to all MET calls
- All EMS calls: We make an Utstein type analyze to all EMS calls during June 2015
- All patient in the emergency department: We make an Utstein type analyze to all Emergency visits during June 2015

SUMMARY:
Patients in general wards have abnormal physical values preceding in-hospital cardiac arrest or a transfer to intensive care unit (ICU). The purpose of Medical Emergency Team (MET) or EMS is to interfere early enough in deteriorating patient status to prevent adverse outcomes like cardiac arrest or transfer to intensive care unit. The aims of this study are to record and analyze the effects of EMS and department of emergency and both afferent and efferent limbs of MET activity in Finnish tertiary Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs or older

Exclusion Criteria:

* under 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult EMS or in-hospital patients with deteriorating vital signs or patients in risk in Tampere University Hospital
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | patients are followed until death

SECONDARY OUTCOMES:
The rates of ICU readmissions | one month to six year
The rates of DNAR orders | one month to six year
The number of patients EMS or medical emergency team is called to treat | one month to six years
  We are going to analyze the number of MET calls and their impact on sudden cardiac arrests in TAUH. The time frame is 1st Jan 2010 -31st Dec 2015. It is known fact that well working MET team inside the hospital should decrease the sudden cardiac arrests. We also analyze the EMS calls and the ED visits in June 2015 to see if patient detoriation is related to sudden in-hospital death.
Patient mortality after 6 mo of discharge | one month to six year
  The patients are followed 6 mo after hospital discharge which has happened in year 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jari Kalliomäki, MD, Principal Investigator — Tampere University Hospital; Sanna Hoppu, MD, PhD, Principal Investigator — Tampere University Hospital; Joonas Tirkkonen, MD, Principal Investigator — Tampere University Hospital; Timo Kontula, MD, Principal Investigator — Tampere University Hospital; Eetu Loisa, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland